CLINICAL TRIAL: NCT06368479
Title: A Prospective Cross-Sectional Study to Evaluate Diagnostic Sensitivity and Specificity of iStatis HBsAg Test at the Point-Of-Care Site Settings
Brief Title: Diagnostic Sensitivity and Specificity of iStatis HBsAg Test at the Point-Of-Care Site Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: bioLytical Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: CLS-016B
Record Dates: First submitted 2024-04-10; First posted 2024-04-16 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Hepatitis B; Hepatitis B Infection
Keywords: Hepatitis B rapid test; Hepatitis B infection; Hepatitis B iStatis test; Hepatitis B point of care test
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- iStatis Testing Onsite (Experimental): Capillary (fingerstick) blood samples are tested using iStatis HBsAg Test onsite.
  Interventions: Device: iStatis HBsAg Test
- iStatis Testing In Lab (Experimental): Venous whole blood collected in Ethylenediaminetetraacetic acid tube, plasma and serum samples are tested using iStatis HBsAg Test
  Interventions: Device: iStatis HBsAg Test
- Reference Test (No Intervention): Either serum or plasma sample will be tested on Abbott Architect HBsAg Qualitative Confirmatory Assay and ADVIA Centaur (depending on the test result outcome).

INTERVENTIONS:
Device: iStatis HBsAg Test — Capillary (fingerstick) blood, EDTA venous whole blood, serum and plasma samples to be tested on the iStatis HBsAg Test at the point of care setting.
  Arms: iStatis Testing In Lab; iStatis Testing Onsite

SUMMARY:
A prospective cross-sectional study in which surgically non-invasive sample-taking is done only for the purpose of testing the samples on iStatis HBsAg Test at the point of care.

DETAILED DESCRIPTION:
Participants are prospctively recruited and enrolled to participate in the study. The Capillary (fingerstick) whole blood, and venous whole blood samples (in serum separating tube (SST) and Ethylenediaminetetraacetic acid (EDTA) tube) are collected by a healthcare professional. Serum and plasma samples will be extracted through laboratory processing of the collected serum separating tube and Ethylenediaminetetraacetic acid VWB, respectively. The collected samples of capillary will be tested on iStatis HBsAg Test. The collected Ethylenediaminetetraacetic acid and serum separating tube VWB will be shipped to the central laboratory to appropriately process and extract serum and plasma samples. Ethylenediaminetetraacetic acid VWB, plasma and serum will be tested on iStatis HBsAg Test in the laboratory. An aliquot of the obtained plasma sample will be further tested for reference and confirmatory testing.

The results from iStatis HBsAg Test results will not be used for participant management decisions.

ELIGIBILITY:
Inclusion Criteria:

* Participants/subjects (males, females, and pregnant women) getting tested for Hepatitis B virus for one or more of the following reasons:

  * at risk for Hepatitis B virus
  * having signs and symptoms indicative for Hepatitis B virus
  * Routine testing Unknown or other reasons will be captured
* Participants/subjects of 18 years or older and, who are able to give/sign the informed consent.

Exclusion Criteria:

* Participant younger than 18 years old
* Participants unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Actual)
Dates: Start 2024-03-19 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2024-07-19 (Actual)

PRIMARY OUTCOMES:
iStatis Performance | 3 Months
  To evaluate the device performance i.e. diagnostic sensitivity and diagnostic specificity of the iStatis Hepatitis B surface Antigen (HBsAg) Test compared to comparator assay.

CONTACTS AND LOCATIONS:
Locations (1):
- Epicentre Health Research, Hillcrest, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: No